CLINICAL TRIAL: NCT06135519
Title: Dermogenesis With Mesenchymal Stem Cells: A Fabulous Remedy For Post Acne Depressed Spots
Brief Title: Dermogenesis With Mesenchymal Stem Cells
Acronym: MSCs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Afzaal Bajwa, Assistant Professor, King Edward Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kemu/23/2
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Dermal Regeneration

STUDY DESIGN:
Intervention Model Description: Group A with MSCs Group B with Fat
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cells (Experimental): Mesenchymal Stem Cells taken from adipose tissue will be used
  Interventions: Procedure: Autologous Mesenchymal stem cells injection
- Homogenized fat (Experimental): Adipose tissue will be harvested and used
  Interventions: Procedure: Homogenized fat injection

INTERVENTIONS:
Procedure: Autologous Mesenchymal stem cells injection — Autologous Mesenchymal stem cells will be seperated from harvested fat and injected in acne scars
  Arms: Mesenchymal stem cells
Procedure: Homogenized fat injection — Autologous fat will be harvested, homogenized and injected.
  Arms: Homogenized fat

SUMMARY:
Dermogenesis With Mesenchymal Stem Cells in treating Post Acne Depressed Spots

DETAILED DESCRIPTION:
management at two different stages of the course of the disease. First one at the stage of active disease which needs cleansers, antibiotics, retinoids, anti inflammatory agents and hormonal manipulation. Once active disease is over, patients report to clinician with depressed spots which are caused by localized dermal disruption and fat atrophy post inflammation or spontaneous epithelial rupture or scratching by the patient. These acne spots are hard to treat due to many reasons. Firstly, excision is difficult as size of most of them is small and they are in a large in number. Secondly, filling with and without subcision is not adequately addressing the deformity. Currently, a combination of filling with synthetic filler or fat and resurfacing by peeling, LASER or dermabrasion is in practice. In-spite of all, a treatment is still required to address post acne spots (Ice Spec Spots) adequately.

ELIGIBILITY:
Inclusion Criteria:

* Acne spots

Exclusion Criteria:

* Active acne

Max Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-23 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Dermal thickness | 3 months
  on microscopy of biopsy section

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Cumulative ananlysis

REFERENCES:
- [Derived] Bashir A, Choudhery MS, Afzaal S, Ali S, Afzaal S. Adipose Tissue-Derived Stem Cells Enhance Dermogenesis of Post-Acne Depressed Spots. J Cosmet Dermatol. 2025 Oct;24(10):e70399. doi: 10.1111/jocd.70399. PMID 41078325